CLINICAL TRIAL: NCT06866834
Title: Examination of the Effect of Nocturia on Pelvic Floor Symptoms, Chronotype, Sleepiness, Sleep Quality, Fatigue and Quality of Life in Women with Urinary Incontinence
Brief Title: Examination of the Effect of Nocturia on Pelvic Floor Symptoms, Sleep Parameters and Quality of Life in Women with Urinary Incontinence
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Gulhane School of Medicine
Other Study IDs: 2024-556
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Women; Urinary Incontinence (UI); Nocturia
MeSH Terms: conditions — Urinary Incontinence; Nocturia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group with nocturia: Women who experience urinary incontinence and have nocturia.
- Group without nocturia: Women who experience urinary incontinence but do not have nocturia.

SUMMARY:
Urinary incontinence (UI), a common issue, is the involuntary leakage of urine that negatively affects individuals socially, physically, and psychologically, leading to a decreased quality of life. Nocturia, which is often seen alongside UI, has similar adverse effects. Nocturia refers to the number of urinations during the main sleep period, and it should be accompanied by the intention to fall back asleep after waking up. Nocturia can arise from factors such as sleep disorders and circadian rhythm disturbances. The circadian rhythm regulates the body's biological functions, and this rhythm varies from person to person, creating chronotypes. There is a strong relationship between sleep and nocturia because nocturia leads to deep sleep loss, an increased risk of metabolic diseases, decreased sleep quality and sleep efficiency, and an increase in the number of awakenings after sleep onset. It is necessary to distinguish whether nocturia, which has a comprehensive impact, affects pelvic floor symptoms, chronotype, sleep quality, fatigue, sleepiness, and quality of life in women with UI. Therefore, the aim of this study is to examine the effect of nocturia on pelvic floor symptoms, chronotype, sleepiness, sleep quality, fatigue, and quality of life in women with UI.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is defined as the involuntary leakage of urine. UI, which is commonly observed both globally and in our country, negatively affects individuals socially, physically, and psychologically, decreasing their quality of life. Nocturia, which is frequently seen alongside UI, has similar adverse effects. Nocturia is defined as the number of urinations during the main sleep period, and for these urinations to be considered as nocturia, the intention to fall back asleep after waking must be present. Nocturia can result from various causes, such as sleep disorders and circadian rhythm disturbances. Sleep is one of the biological functions regulated by the 24-hour cycle of body temperature, hormonal balance, hunger and satiety, cognitive and physical performance. This rhythm varies from person to person and creates chronotypes. Based on these chronotypes, the time during the day when individuals function best and when circadian time is regulated differs. There is an undeniable relationship between sleep and nocturia. Nocturia causes loss of deep sleep, known as slow-wave sleep, increases the risk of metabolic diseases, decreases sleep quality and sleep efficiency, and increases the number of awakenings after sleep onset. This decrease in sleep quality can lead to increased sleepiness, fatigue, and reduced quality of life. It is necessary to differentiate whether nocturia, which has a comprehensive effect, influences pelvic floor symptoms, chronotype, sleep quality, fatigue, sleepiness, and quality of life in women with UI. Therefore, the aim of this study is to investigate the effect of nocturia on pelvic floor symptoms, chronotype, sleepiness, sleep quality, fatigue, and quality of life in women with UI.

2. Materials and Methods

Participants: Participants in the study will be selected from patients who visit the Gynecology and Obstetrics Outpatient Clinic at GATA Training and Research Hospital. The study will include patients over the age of 18 who experience incontinence. After the patients are informed about the study, written and verbal consent will be obtained from them. The sample size for the study was calculated using the G*Power 3.1 program with a power of 80% and a type 1 error level of 0.05. It was calculated that a total of 102 people, with at least 51 participants in each group (with and without nocturia), would be required. The exclusion criteria for the study include sleep disorders, neurological diseases, chronic kidney disease, the use of sleep medication, antidepressants, diuretics, or urinary incontinence drugs, hormone replacement therapy, pregnancy or childbirth within the last six months, urinary tract infections in the last three months, prolapse beyond stage 2, orthopedic trauma to the pelvic region or pelvic surgery within the last six months, and a history of cancer.

Evaluation: A semi-structured evaluation form will be used to record the demographic data of the participants. The participants' anthropometric features such as age (years), height (cm), weight (kg) will be recorded. Educational level, marital status, occupation, main complaint, and duration of complaints (months) will be queried. Their medical history, surgeries, family history, medications, smoking, chronic cough, and constipation status will be noted. Obstetric history and menstrual status will be collected. The type of incontinence will be evaluated using the 3 Incontinence Questions (3IQ) survey, urinary symptoms will be assessed with the Global Pelvic Floor Distress Inventory and Urogenital Distress Inventory-6, chronotypes will be evaluated using the Morningness-Eveningness Questionnaire, sleepiness will be assessed with the Epworth Sleepiness Scale, sleep quality will be measured using the Pittsburgh Sleep Quality Index, fatigue levels will be evaluated using the Fatigue Severity Scale, and quality of life will be assessed with the CONTILIFE Questionnaire.

3 Incontinence Questions (3IQ): The 3 Incontinence Questions is a simple, repeatable survey used to determine the type of urinary incontinence. It classifies the patient into stress, urge, mixed, or other types based on the most common situation in which they experience urinary leakage over the last three months. The 3 Incontinence Questions is an open-access form that does not require permission for use.

Global Pelvic Floor Distress Inventory and Urogenital Distress Inventory-6: To assess discomfort from symptoms of pelvic floor dysfunction, the Turkish validated Global Pelvic Floor Distress Inventory and Urogenital Distress Inventory-6 will be used. Higher scores on these scales indicate greater severity of discomfort.

Morningness-Eveningness Questionnaire: Participants' chronotype will be evaluated using the Turkish validated Morningness-Eveningness Questionnaire. The questionnaire consists of 19 questions, and the score ranges from 16 to 86. The score can be divided into three ranges, each representing a different chronotype: a score of 59-86 indicates a morning type, 42-58 indicates an intermediate type, and 16-41 indicates an evening type.

Epworth Sleepiness Scale: Participants' daytime sleepiness will be assessed using the Turkish validated Epworth Sleepiness Scale. This scale consists of 8 items, each scored from 0 (never doze) to 3 (high chance of dozing). The higher the score, the greater the level of daytime sleepiness.

Pittsburgh Sleep Quality Index: The Turkish validated Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. PSQI includes seven subcategories that evaluate aspects of sleep such as sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. The total score ranges from 0 to 21, with scores of 5 or below indicating "good" sleep quality, and scores above 5 indicating "poor" sleep quality.

Fatigue Severity Scale: Participants' fatigue severity will be evaluated using the Turkish validated Fatigue Severity Scale. This scale consists of 9 questions, with each question rated on a Likert scale from 1 (strongly disagree) to 7 (strongly agree). The total score is determined by the arithmetic mean of the responses, and a score of 4 or above indicates the presence of fatigue.

CONTILIFE Questionnaire: The CONTILIFE Questionnaire is a quality of life scale specifically developed for urinary incontinence and has been validated in Turkish. It consists of six subparameters related to daily and effort activities, self-image, emotional status, sexuality, and well-being, and contains 28 questions. Each question is rated on a Likert scale from 1 to 5 or 0 to 5, with higher scores indicating better quality of life.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Group with Nocturia:

* Being 18 years of age or older
* Being female
* Have been diagnosed with urinary incontinence
* Wake up during the main sleep period to relieve the need to urinate, with the intention of returning to sleep or falling asleep again after each urination

Inclusion Criteria for the Group without Nocturia:

* Being 18 years of age or older
* Being female
* Have been diagnosed with urinary incontinence

Exclusion Criteria:

Exclusion Criteria for the Group with Nocturia:

* Diagnosis of a sleep disorder
* Diagnosis of any neurological disease
* Chronic kidney disease
* Diagnosis of diabetes
* Use of sleep medications
* Use of antidepressants
* Use of diuretic medications
* Use of any medication for urinary incontinence
* Hormone replacement therapy
* Pregnancy or having given birth within the last six months
* Having had a urinary tract infection in the last three months
* Presence of prolapse greater than stage 2
* History of orthopedic trauma to the pelvic region
* Pelvic surgery within the last six months
* History of cancer

Exclusion Criteria for the Group without Nocturia:

* Waking up during the main sleep period to relieve the need to urinate, with the intention of returning to sleep or falling asleep again after each urination
* Diagnosis of a sleep disorder
* Diagnosis of any neurological disease
* Chronic kidney disease
* Diagnosis of diabetes
* Use of sleep medications
* Use of antidepressants
* Use of diuretic medications
* Use of any medication for urinary incontinence
* Hormone replacement therapy
* Pregnancy or having given birth within the last six months
* Having had a urinary tract infection in the last three months
* Presence of prolapse greater than stage 2
* History of orthopedic trauma to the pelvic region
* Pelvic surgery within the last six months
* History of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Gülhane Training and Research Hospital, Department of Obstetrics and Gynecology
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Symptoms | from January 2025 to April 2025
  To determine the discomfort caused by pelvic floor dysfunction symptoms, the "Global Pelvic Floor Discomfort Questionnaire" will be used.
  The Global Pelvic Floor Discomfort Questionnaire consists of 9 questions. The score obtained from the scale ranges from 0 to 45, and to convert this score to a percentage, the total score is averaged and then multiplied by 20. As the score on the scale increases, the severity of the discomfort also increases.
Assessment of Symptoms | from January 2025 to April 2025
  To determine the discomfort caused by pelvic floor dysfunction symptoms, the "Urogenital Distress Inventory-6" will be used.
  The Urogenital Distress Inventory is a Likert-type scale consisting of 6 questions. The score obtained from the scale ranges from 0 to 18, and the score is converted into a percentage. As the score on the scale increases, the severity of the discomfort also increases.
Assessment of Sleep Quality | from January 2025 to April 2025
  Pittsburgh Sleep Quality Index will be used.Pittsburgh Sleep Quality Index scale has seven sub-scales that portray various domains of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Responses for each subscale are scored as 0-3. Having a global score of 5 or higher indicates bad sleep quality. sleepiness.
Assessment of Chronotype | from January 2025 to April 2025
  Chronotype assessment will be evaluated using the "Morningness-Eveningness Questionnaire." The questionnaire consists of 19 questions. It has a five-point scale, with each range corresponding to a different chronotype. Individuals who score between 70-86 are classified as "definitely morning type," those who score between 59-69 are classified as "closer to morning type," those who score between 42-58 are classified as "intermediate type," those who score between 31-41 are classified as "closer to evening type," and individuals who score between 16-30 are classified as "definitely evening type."
Assessment of Quality of life | from January 2025 to April 2025
  Quality of life will be assessed using the CONTILIFE Questionnaire. The questionnaire is a Likert-type scale consisting of 28 questions and includes six subparameters. Questions 1-7 assess daily activities, questions 8-11 assess effort, questions 12-18 assess self-esteem, questions 19-24 assess emotional impact, questions 25-27 assess sexuality, the 28th question is used to evaluate general quality of life.The total score is determined by summing the scores from all subparameters. As the total score increases, it indicates a poorer quality of life.

SECONDARY OUTCOMES:
Assessment of Sleepiness | from January 2025 to April 2025
  Epworth Sleepiness Scale(ESS) will be used. Its score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime
Assessment of Fatigue | from January 2025 to April 2025
  Fatigue will be assessed using the Fatigue Severity Scale (FSS). The FSS consists of 9 items designed to evaluate the severity of fatigue and its impact on daily activities. Each item is scored on a 7-point Likert scale, where 1 represents "strongly disagree" and 7 represents "strongly agree." Higher scores indicate greater fatigue severity. The total score is calculated by averaging the responses across all items. Scores of 4 or above indicate the presence of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Physiotherapy and Rehabilitation, Ankara, Keçiören, Turkey (Türkiye)